CLINICAL TRIAL: NCT04846478
Title: A Phase Ia/Ib Study of Talazoparib in Combination With Tazemetostat in Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Phase Ia/Ib Talazoparib + Tazemetostat for mCRPC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Epizyme, Inc. (Industry); Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Atish Choudhury, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-086
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — talazoparib; tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Talazoparib + Tazemetostat (Experimental): Standard 3+3 dose escalation will be followed, participants will initially receive talazoparib and tazemetostat at a dose of 75% of the starting dose for their FDA-approved indications.
  During each 28 day study treatment cycle participants will take:
  * Talazoparib once daily.
  * Tazemetostat twice daily.
  Interventions: Drug: Talazoparib; Drug: Tazemetostat
- Dose Expansion Talazoparib + Tazemetostat (Experimental): Participants will receive talazoparib and tazemetostat at the safe dose identified in the first part (dose escalation) of the study.
  During each 28 day study treatment cycle participants will take:
  * Talazoparib once daily.
  * Tazemetostat twice daily.
  Interventions: Drug: Talazoparib; Drug: Tazemetostat

INTERVENTIONS:
Drug: Talazoparib — capsule, taken by mouth, once a day
  Other Names: Talzenna
Drug: Tazemetostat — orally as a tablet twice daily.
  Other Names: Tazverik; EPZ-6438

SUMMARY:
This trial is testing whether molecularly targeted oral medications called talazoparib and tazemetostat can be safely combined for the treatment of prostate cancer, and whether the combination is effective in shrinking or preventing the growth of metastatic prostate cancer.

The names of the study drugs involved in this study are:

* Talazoparib
* Tazemetostat

DETAILED DESCRIPTION:
This is a Phase 1a/1b clinical trial to assess safety, tolerability and preliminary clinical activity of the combination of talazoparib with tazemetostat in metastatic castration-resistant prostate cancer (mCRPC) patients.

The U.S. Food and Drug Administration (FDA) has not approved talazoparib or tazemetostat for metastatic castration-resistant prostate cancer (mCRPC) but they have been approved for other uses. Talazoparib has been approved for use in breast cancer, and tazemetostat has been approved for use in certain types of sarcoma and lymphoma.

Talazoparib is an orally administered molecularly targeted chemotherapy drug called a "PARP inhibitor", which acts to block the ability of cancer cells to repair certain forms of damage to their DNA - the accumulation of damaged DNA causes certain cancer cells to die. Other PARP inhibitors are already approved for use in prostate cancer patients with specific gene mutations detected in their blood or in their cancer, and talazoparib is currently being studied for treatment of prostate cancer in other clinical trials.

Tazemetostat is an orally administered molecularly targeted chemotherapy drug called an "EZH2 inhibitor", which acts to block the production of proteins encoded by DNA in the cancer cells that are important in cancer growth and survival. Tazemetostat is also being studied for the treatment of prostate cancer in other clinical trials. In the laboratory setting, tazemetostat causes changes in protein levels in prostate cancer cells that make them sensitive to dying in the presence of PARP inhibitors.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

The study design involves two parts. The first part is called the "dose escalation" to find a safe dose for the combination of talazoparib and tazemetostat. The second part is called the "dose expansion" where additional participants are treated at the safe dose identified in the first part of the study.

Participants will receive study treatment for as long as they do not have serious side effects and their disease does not get worse. Participants will be followed after completion of study treatment for up to 24 months.

It is expected that about 38 people will take part in this research study.

Funding for this research is provided by a grant awarded by the non-profit Prostate Cancer Foundation along with Pfizer, Inc. In addition, Pfizer is supporting the study by providing the study drug talazoparib. Epizyme, Inc. is supporting the study by providing the study drug tazemetostat.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate cancer (code 10036910) with progressive disease at the time of study entry by either

  * Sequence of at least 2 rising PSA values at a minimum of 1-week intervals
  * Radiographic progression per RECIST1.1 for soft tissue and/or per PCWG3 for bone, with or without PSA progression
* Patients must have metastatic disease by bone scintigraphy or other nodal or visceral lesions on CT or MRI with a bone or soft tissue lesion amenable to image-guided percutaneous biopsy, a castrate level of testosterone (<50ng/dL), and evaluable for disease response by either

  * Baseline PSA ≥ 2.0 ng/mL OR
  * Measurable disease per RECIST 1.1 NOTE: Subjects must maintain a castrate state. If they have not had an orchiectomy, they must continue to receive LHRH or GnRH agonists or antagonists unless intolerant.
* Past progression on at least one novel hormonal therapy (abiraterone, enzalutamide, apalutamide, darolutamide, galeterone, orteronel, seviteronel or equivalent) in either the hormone-sensitive or castration-resistant disease setting.
* Not a candidate for docetaxel or cabazitaxel chemotherapy due to:

  * progression within 12 months of completion or intolerance to prior taxane OR
  * refusal of taxane OR
  * contraindication to, or lack of fitness for taxane OR
  * investigator assessment that taxane is not clinically indicated or preferred
* Age ≥18 years. Children under 18 are excluded from this study as prostate cancer is a disease of adults
* ECOG performance status ≤1 (Karnofsky ≥70%, see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * hemoglobin ≥9 g/dL (without transfusion or growth factor in prior 28 days)
  * platelets ≥ 100,000/mcL (without transfusion of growth factor in prior 28 days)
  * total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) unless known or suspected Gilbert syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 (based on Cockcroft-Gault formula OR creatinine clearance based on 24 hour urine collection)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy (with no known or predicted drug-drug interactions with talazoparib and/or tazemetostat) with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable. If suppressive therapy is indicated, there must be no known or predicted drug-drug interactions with talazoparib and/or tazemetostat.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if there are no known or predicted drug-drug interactions with talazoparib and/or tazemetostat and they have an undetectable HCV viral load.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Prior treatment with a PARP inhibitor is allowed.
* Planned to undergo core biopsy of a recurrent/metastatic lesion adequate for next generation sequencing (NGS) after trial registration but prior to cycle 1 day 1 of therapy. Confirmation of adequacy of this biopsy material for NGS is NOT required for initiation of therapy. If elective biopsies are not being performed at the treating institution due to preparations or precautions related to COVID-19, this requirement can be waived on discussion with the trial PI.
* Willing to undergo core biopsy of a recurrent/metastatic lesion adequate for next generation sequencing (NGS) after 8 weeks (+/- 7 days) of study treatment.
* The effects of talazoparib and tazemetostat on the developing human fetus are unknown. For this reason and because oral chemotherapeutic agents are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of talazoparib and tazemetostat administration.
* Ability to swallow oral medications.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy, intravenous experimental agent, radiopharmaceutical therapy or radiotherapy within 4 weeks prior to planned cycle 1 day 1 of study treatment.
* Participants who have received oral anti-neoplastic intervention such as an oral hormonal agent, PARP inhibitor, or oral experimental agent within 14 days prior to planned cycle 1 day 1 of study treatment.
* Participants who have not recovered from clinically significant adverse events due to prior anti-cancer therapy (i.e., have clinically significant residual toxicities > Grade 1) except for stable complications of prior procedures (such as urinary incontinence or erectile dysfunction) or Grade 2 anorexia, alopecia, neuropathy, and fatigue, for which resolution is not required.
* Participants who are receiving any other investigational agents.
* Participants previously treated with an inhibitor of EZH2.
* Patients with known brain metastases or leptomeningeal disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talazoparib or tazemetostat.
* Participants receiving the following concurrent medications:

  * Participants receiving the P-gp inhibitors amiodarone, carvedilol, clarithromycin, itraconazole, or verapamil are ineligible. Participants receiving other P-gp inhibitors are not excluded but should be monitored for potential increased adverse reactions.
  * Participants receiving BCRP inhibitors are not excluded but should be monitored for potential increased adverse reactions.
  * Participants receiving any medications or substances that are strong or moderate inhibitors or inducers of CYP3A4 are ineligible.
  * Precaution is warranted with concomitant use of agents with a narrow therapeutic index that are substrates of CYP3A4 and/or P-gp.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

* Participants with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded from this study because they do not develop prostate cancer.
* Arterial or venous thromboembolic event within the last 3 months.
* Concurrent active malignancy. Patients with non-melanomatous skin cancer, superficial bladder cancer, cancer not needing active therapy for at least 2 years, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are also permitted to enroll.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Dose Limiting Toxicity (DLT) | Enrollment up to 28 days
  Assessed by the investigator, based on toxicity grade (according to the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0), clinical significance, and possible relationship to either study drug.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | Enrollment up to 2 years
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Enrollment up to 2 years
  Assessed by RECIST 1.1 and/or prostate-specific antigen (PSA) reduction by ≥ 50%

CONTACTS AND LOCATIONS:
Overall Officials: Atish Choudhury, MD PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu